CLINICAL TRIAL: NCT00785044
Title: An Open-label, Multicentre, Phase 3 Study to Demonstrate the Prognostic Usefulness of 123I-mIBG Scintigraphy for Identifying Subjects With Heart Failure Who Will Experience an Adverse Cardiac Event During 24 Months Followup
Brief Title: Study Dosed With (123I-mIBG) for Identifying Subjects With Heart Failure Who Will Experience an Adverse Cardiac Event
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: MBG313
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Congestive Heart Failure
Keywords: Heart Failure; MIBG; 123I-mIBG
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group: No participants received any drug administration. No intervention conducted.
  Interventions: Drug: I-123 mIBG

INTERVENTIONS:
Drug: I-123 mIBG — This was an observational study. Participants were previously dosed in separate study.

SUMMARY:
The study was designed to study the utility of meta-iodobenzylguanidine (123I-mIBG) imaging to identify those participants with heart failure who would experience an adverse cardiac event during 24 months of follow-up from the administration date of 123I-mIBG in previous studies MBG311 or MBG312.

ELIGIBILITY:
Inclusion Criteria:

* The subject was a Heart Failure subject who signed informed consent for MBG311, MBG312, or MBG312C.
* The subject was administered 123I-mIBG in MBG311, MBG312, or MBG312C.
* The subject completed the late planar imaging assessments (at a minimum) required by the protocols for MBG311, MBG312, or MBG312C.
* The subject agreed to allow the investigator access to medical records, including those relating to subject death should this occur.

Exclusion Criteria:

* The subject withdrew or was withdrawn from MBG311, MBG312, or MBG312C.
* The subject was considered lost-to-follow-up (6 months without contact) in MBG311, MBG312, or MBG312C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure Participants who participated in: MBG311 (NCT00126425) and MBG312/312C (NCT00126438).
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Strohmeyer, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the present study MBG313 (NCT00785044), participants previously administered AdreView™ (123I-mIBG [meta-iodobenzylguanidine]) in studies MBG311 (NCT00126425) and MBG312 (NCT00126438) were monitored for up to 24 months from the date of administration of 123I-mIBG.
Pre-assignment Details: Of 964 heart failure (HF) participants included in efficacy population of MBG311 (NCT00126425) and MBG312 (NCT00126438), 471 participants signed informed consent and enrolled into extension MBG313 study and provided additional efficacy data. New data from MBG313 study combined with data collected in MBG311 and MBG312 studies for efficacy analysis.
Groups:
- AdreView™- Heart Failure Group: HF participants administered AdreView™ (123I-mIBG [meta-iodobenzylguanidine]) in studies MBG311 (NCT00126425) and MBG312 (NCT00126438) were monitored for up to 24 months at 6-month intervals from the date of administration of 123I-mIBG to assess the occurrence of adverse cardiac events (ACEs).
Period: Overall Study
Arm/Group | AdreView™- Heart Failure Group
Started | 964 (Eligible to participate in MBG313)
Enrolled Participants | 471 (Out of 964 from MBG311 and MBG312 HF participants, 471 enrolled into the extension MBG313 study.)
Completed | 468 (Data for 471 participants (MBG313) combined with data from MBG311 and MBG312 for efficacy analysis)
Not Completed | 496
Not completed — Dosed at non-participating sites | 152
Not completed — Death | 77
Not completed — Lost to Follow-up | 266
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- AdreView™ - Heart Failure Group: HF participants administered AdreView™ (123I-mIBG [meta-iodobenzylguanidine]) in studies MBG311 (NCT00126425) and MBG312 (NCT00126438) were monitored for up to 24 months at 6-month intervals from the date of administration of 123I-mIBG to assess the occurrence of ACEs.
Arm/Group | AdreView™ - Heart Failure Group
Number analyzed (Participants) | 964
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192
  Male | 772

OUTCOME MEASURES:

1. Primary Outcome: Numerical Heart to Mediastinum (H/M) Ratio at 3 Hours 50 Minutes Post-administration on Planar 123I-mIBG Imaging by Adverse Cardiac Events (ACEs) Status
Description: The numerical value of 123 I-mIBG uptake (H/M ratio) at 3 hours 50 minutes post administration was calculated by dividing the counts/pixel in the total myocardium region of interest (ROI) by the counts/pixel in the 7x7 pixel mediastinal ROI. Receiver operator characteristic curves (ROC) constructed on the basis of sensitivity and specificity to identify ACEs across all H/M values were used to calculate the area under the ROC curve (AUC). The AUC was used to test for statistical significance of the prognostic usefulness of the H/M ratio. In the present MBG313 study, additional efficacy data is provided for 471 participants and new data from MBG313 were combined with data collected in MBG311 and MBG312 for efficacy analysis.
Time Frame: From the date of administration of 123I-mIBG in studies MBG-311 or MBG-312 up to 24 months
Population: Efficacy population was 961 participants who received IMP and had a consensus H/M ratio on 3 hour 50 minute planar image in MBG 311 or MBG 312. Here, number of participant analyzed = number of participants with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- AdreView™ - HF Group (With No Adverse Cardiac Events): HF participants administered AdreView™ (123I-mIBG [meta-iodobenzylguanidine]) in studies MBG311 (NCT00126425) and MBG312 (NCT00126438) with no ACEs monitored for up to 24 months at 6-month intervals from the date of administration of 123I-mIBG.
- AdreView™- HF Group (With Adverse Cardiac Events): HF participants administered AdreView™ (123I-mIBG [meta-iodobenzylguanidine]) in studies MBG311 (NCT00126425) and MBG312 (NCT00126438) with ACEs monitored for up to 24 months at 6-month intervals from the date of administration of 123I-mIBG.
Arm/Group | AdreView™ - HF Group (With No Adverse Cardiac Events) | AdreView™- HF Group (With Adverse Cardiac Events)
Number analyzed (Participants) | 829 | 132
Ratio | 1.451 (0.2033) | 1.394 (0.1885)
Statistical Analysis 1: Comparison: AdreView™ - HF Group (With No Adverse Cardiac Events) vs AdreView™- HF Group (With Adverse Cardiac Events); Analysis was performed on all HF participants from both groups "AdreView™ - HF Group (With No Adverse Cardiac Events)" and "AdreView™ - HF Group (With Adverse Cardiac Events)" based on H/M ratio; Test type: Superiority or Other — Analysis was performed using the null hypothesis for the AUC stated as: H0: θ ≤A versus H1: θ >A, where the AUC (θ) value was: 'A' selected based on the diagnostic utility desired from the use of myocardial 123 I-mIBG uptake measured using H/M ratio. A smooth parametric model of the ROC curve was fitted to the data. The AUC for the resulting model was calculated and 95% confidence interval for the AUC was reported. The hypothesis was tested using the Z-statistics at 'A' at level of 0.70; p < 0.001, Z-statistic — At 0.05 level of significance; Mean = 0.581, 95% CI 2-sided [0.532 to 0.630]

ADVERSE EVENTS:
Description: The main objective of the study was to monitor participants previously administered AdreView™ (123I-mIBG [meta-iodobenzylguanidine]) in studies MBG311 (NCT00126425) and MBG312 (NCT00126438) to identify participants at higher risk of experiencing an adverse cardiac event up to 24 months from the date of administration of 123I-mIBG, therefore, no safety evaluations performed in this study.
Arm/Group | AdreView™ - Heart Failure Group
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Designed as a continuation of original phase 3, but objectives were built around analyses of integrated data from both studies. Distinct from endpoints used in MBG311 and MBG312. No intent to analyze current study on single original study basis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.